CLINICAL TRIAL: NCT01048268
Title: Glucose-dependent Insulinotropic Polypeptide - New Role as Blood Glucose Stabilizer?
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Mikkel Christensen, MD, PhD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GIP HYPO (MC)
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes Mellitus
Keywords: T1DM; T2DM; GIP; Glucose-dependent insulinotropic polypeptide; Incretin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Incretins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy volunteers (Experimental)
  Interventions: Drug: glucose-dependent insulinotropic polypeptide; Drug: Placebo
- Patients with Type 1 diabetes mellitus (Experimental)
  Interventions: Drug: glucose-dependent insulinotropic polypeptide; Drug: Placebo
- Patients with type 2 diabetes mellitus (Experimental)
  Interventions: Drug: glucose-dependent insulinotropic polypeptide; Drug: Placebo

INTERVENTIONS:
Drug: glucose-dependent insulinotropic polypeptide — For the first 20 min of the experiment the volunteers will receive GIP at 4 pmol/kg body weight.
  For the following 40 minutes the volunteers will receive 2 pmol/kg body weight
Drug: Placebo — copy GIP infusion rates

SUMMARY:
The purpose of this study is to determine whether glucose-dependent insulinotropic polypeptide (GIP) has a stabilizing function on the blood glucose

DETAILED DESCRIPTION:
The aim of the study is to investigate the effect of GIP on the glucagon secretion during hyper-, eu- and hypoglycemia in healthy volunteers, patients with type 1 diabetes mellitus and patients with type 2 diabetes mellitus.

From this, we will evaluate GIP's role as blood sugar stabilizer.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians with T1DM (diagnosed according to WHO's criteria) without residual beta cell function (arginine test without increase in c-peptide) in treatment with long acting insulin OR
* Caucasians with non-insulin treated T2DM (diagnosed according to WHO's criteria) OR
* Caucasians without first degree relative with diabetes mellitus, with normal fasting plasma glucose and glucose tolerance along with negative islet and GAD-65 autoantibodies AND
* Normal hemoglobin
* Informed consent

Exclusion criteria:

* Unwillingness to participate or the wish to leave the present study
* HbA1c > 9 %
* Liver disease (ALAT or ASAT > 2 times normal value)
* Diabetic nephropathy (serum creatinin > 130 microM and/or albuminury)
* Proliferative diabetic retinopathy (anamnetic)
* Atherosclerotic heart disease or heart failure (NYHA group III and IV)
* Anemia
* Treatment with medicine which cannot be paused for 12 hours
* Pregnancy and/or breast feeding
* Fasting plasma glucose > 15 mM on the day of the experiment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The difference in glucagon secretion quantified as the difference in plasma glucagon concentration and incremental baseline-subtracted area under the curve (AUC) for plasma glucagon | -10, 0, 5, 10, 20, 30, 45, 60 and 90 minutes at each visit

SECONDARY OUTCOMES:
The difference between the amount of infused glucose and the insulin responses | will be measured at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel Christensen, MD, Principal Investigator — Bispebjerg Hospital, Copenhagen; Filip K Knop, MD PhD, Study Director — Diabetes Research Division, Department of Internal Medicine F, Gentofte Hospital, University of Copenhagen
Locations (1):
- Department of Internal Medicine F' laboratory, Hellerup, Copenhagen County, Denmark

REFERENCES:
- [Derived] Veedfald S, Vedtofte L, Skov-Jeppesen K, Deacon CF, Hartmann B, Vilsboll T, Knop FK, Christensen MB, Holst JJ. Glucose-Dependent Insulinotropic Polypeptide Is a Pancreatic Polypeptide Secretagogue in Humans. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgz097. doi: 10.1210/clinem/dgz097. PMID 31665480